CLINICAL TRIAL: NCT00225030
Title: Observational Study of the Prognosis in Treated Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Other Study IDs: SHAP-DK
Record Dates: First submitted 2005-09-13; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2004-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

INTERVENTIONS:
Drug: antihypertensive drugs according to current guidelines

SUMMARY:
Observational study of life time prognosis for persons medically treated for arterial hypertension, according to current WHO-guidelines.

ELIGIBILITY:
Inclusion Criteria:

hypertension according to WHO-defined criteria

Exclusion Criteria:

age < 18 years

pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 1970-01; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Michael Strate, MD, Principal Investigator
Locations (1):
- Medicial Dept. C, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Result] Strate M, Vaeth M, Harvald B. Twenty-one-year survival of primary hypertensive patients allocated to care in general practice or in specialized hypertension clinic. An observational study of 831 hypertensive patients. Blood Press. 1997 Mar;6(2):88-95. doi: 10.3109/08037059709061805. PMID 9105647